CLINICAL TRIAL: NCT05711550
Title: Investigating the Effect of Normal Frequency-band and Infra-low Frequency Neurofeedback on Functional Brain Connectome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipp Stämpfli (Other)
Responsible Party: Sponsor-Investigator, Philipp Stämpfli, Head of MR Center, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ILF_NFB_Allstudies
Record Dates: First submitted 2023-01-13; First posted 2023-02-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Neurofeedback
Keywords: Neurofeedback, fMRI, resting-state

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Subjects: Study 1 (Experimental): This arm corresponds to study 1 (Real Neurofeedback uses only normal frequency band signals ranging from 1 to 35 Hz from the EEG-signal). All included participants participate at 2 experimental conditions (Real Neurofeedback, Sham Neurofeedback) at 2 different days in a randomized order. Both, the investigators and the participants are blinded in regard to the intervention they receive at the two experimental visits.
  Interventions: Device: Real Neurofeedback; Device: Sham Neurofeedback
- Healthy Subjects: Study 2 (Experimental): This arm corresponds to study 2 (Real Neurofeedback uses only infra-low frequencies below 0.1Hz from the EEG-signal). All included participants participate at 2 experimental conditions (Real Neurofeedback, Sham Neurofeedback) at 2 different days in a randomized order. Both, the investigators and the participants are blinded in regard to the intervention they receive at the two experimental visits.
  Interventions: Device: Real Neurofeedback; Device: Sham Neurofeedback
- Healthy Subjects: Study 3 (Experimental): This arm corresponds to study 3 (normal frequency band & infra-low frequencies are used in Real Neurofeedback). All included participants participate at 2 experimental conditions (Real Neurofeedback, Sham Neurofeedback) at 2 different days in a randomized order. Both, the investigators and the participants are blinded in regard to the intervention they receive at the two experimental visits.
  Interventions: Device: Real Neurofeedback; Device: Sham Neurofeedback

INTERVENTIONS:
Device: Real Neurofeedback — Real Neurofeedback with visual and acoustic feedback presentation based on the EEG-signal from the participant (Signals used described in corresponding study arm). The NFB-signals are obtained from the T4 and P4 positions according to the 10-20 EEG placement consensus. NFB is done using the software package Cygnet (BEE Medic GmbH Technologies, Kirchberg, Switzerland) and for all participants the same neurofeedback-animation is used. NFB training duration is approx. 30min
Device: Sham Neurofeedback — The sham neurofeedback is performed in identical fashion using the same software, feedback, electrode placement, duration as in the real neurofeedback. Only difference is that a pre-recorded EEG-dataset will be used and the feedback signal is thus independent from the brain activity of the participant.

SUMMARY:
In this basic research project a novel form of neurofeedback is investigated, in which in addition to the use of 1) normal frequency bands (1-35 Hertz), 2) very slow signals (low frequency; < 0.1 Hertz) are used, which correspond more to the basic excitability of the brain. Because of the slow signal characteristics, this method is called infra-low frequency neurofeedback (ILF-NFB for short). Although this method has been successfully applied in clinical settings since the 1980s, the mechanisms underlying the effect are largely unexplored. For that purpose, a project consistiong of three studies will be conducted in order to investigate the neurophysiological effects of both signal elements on healthy participants:

* Study 1 examines the effects of normal frequency band training alone.
* Study 2 examines the effects of low frequency training.
* Study 3 examines the effects of the combination of normal frequency band and low frequency training

For each study, a total of 40 clean data sets are to be collected, resulting in a minimum amount of 120 participants for all three studies.

All three studies investigate the effects of the neurofeedback on brain connectivity patterns by means of functional magnetic resonance imaging (fMRI), accompanied by measurements of the autonomic nervous system (ANS) and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Written informed consent after participants' information
* Fluent in German language (required for an adequate answering of the questionnaires)
* No previous experience with neurofeedback treatments

Exclusion Criteria:

* Alcohol, drug and analgesics consumption within the last 24 hours
* Pre-existing neurological and/or psychiatric conditions
* History of brain injuries
* Alcohol and drug abuse
* Chronic diseases that require permanent medication
* Exclusion criteria met based on the screening questionnaire
* General contraindications for MR-testings (e.g. claustrophobia, pace maker, cochlear implant, insulin pump)
* Hypersensitivity to loud noises
* Incapable of lying still during a longer period of time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Functional brain connectivity | 90 Minutes
  Comparison of the Pre-Post intervention differences in resting state functional connectivity (assessed using fMRI)

SECONDARY OUTCOMES:
Heart rate Variability Pre/Post Interventions | 90 Minutes
  Comparison of the Pre-Post intervention differences in heart rate variability (during fMRI measurements)
Respiration frequency Pre/Post Interventions | 90 Minutes
  Comparison of the Pre-Post intervention differences in respiration frequency (during fMRI measurements)
Heart rate variability during interventions | 30 Minutes
  Comparison of heart rate variability measured during both interventions (Neurofeedback and Sham Neurofeedback)
Respiration frequency during interventions | 30 Minutes
  Comparison of respirateion frequency measured during both interventions (Neurofeedback and Sham Neurofeedback)
Electrodermal activity during interventions | 30 Minutes
  Comparison of electrodermal activity (skin conductance) measured during both interventions (Neurofeedback and Sham Neurofeedback)
Power spectrum density (PSD) of the delta, theta, alpha, beta and gamma bands in the EEG-signal recorded during interventions | 30 Minutes
  Comparison of power spectral density (PSD) of the delta, theta, alpha, beta and gamma frequency bands recorded by the neurofeedback equipment during both interventions (Neurofeedback and Sham Neurofeedback)
Power spectrum density (PSD) of low-frequency components (< 0.1Hz) in the EEG-signal recorded during interventions | 30 Minutes
  Comparison of power spectral density (PSD) of low-frequency components (< 0.1Hz) recorded by the neurofeedback equipment during both interventions (Neurofeedback and Sham Neurofeedback)

OTHER OUTCOMES:
Mental state pre/post intervention | 40 Minutes
  Participants complete a questionnaire immediately before and after intervention for assessment of participants' mental state pre and immediately after the interventions
Sleep questionnaire | 24 Hours
  Questionnaires on sleep quality will be given to the participants at the beginning of each experimental visit and within 24 hours after participation in order to assess effects of the interventions on sleep quality.
Personality questionnaires | 10 Minutes
  BFI-60 personality questionnaire will be completed by participants at the beginning of each experimental visit to assess interactions between personality attributes and other outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Stämpfli, PD PhD, Principal Investigator — Psychiatric University Hospital, Zurich
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided